CLINICAL TRIAL: NCT06180538
Title: EPIVIEWS: Exploring Patient Impact & Value in Epilepsy Wearables for Seizure Monitoring
Brief Title: Exploring Patient Impact & Value in Epilepsy Wearables for Seizure Monitoring
Acronym: EPIVIEWS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EPIVIEWS
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
Keywords: wearable device
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study Is to determine the accuracy and reliability of the wearable device in a controlled environment. This study will inform patients, healthcare professionals, and the wider community of the accuracy of the device in detecting seizures.

DETAILED DESCRIPTION:
Epilepsy is a common serious neurological disorder, regularly presenting with seizures that can affect patients without warning. Any seizure has the potential to cause significant injury to patients or sudden unexplained death in epilepsy (SUDEP). As such, many patients with epilepsy and their caregivers live with a fear that a seizure may occur, fundamentally impacting their quality of life.

New technology including the use of wearable devices have the potential to identify a seizure and notify caregivers immediately of a person in danger. These devices use sensors that look out for the types of movements demonstrated during a seizure and are able to send alerts automatically when connected to a smartphone and the internet. One example of this device is the Empatica Embrace2 which is a wrist worn wearable that has been approved for use in epilepsy. This relatively new technology is available to purchase by the public, but it is not yet clear what value this device offers.

Whilst man of these devices may be been cleared for use by regulators and available to buy on the consumer market. It remains unclear on the value that they can offer to patients. The purpose of this research study Is to determine the accuracy and reliability of the wearable device in a controlled environment. This study will inform patients, healthcare professionals, and the wider community of the accuracy of the device in detecting seizures.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is over the age of 18
2. The participant has access to a smartphone
3. The participant has a history of generalised tonic-clonic seizures in the past year

Exclusion Criteria:

1. The participant lacks capacity to give informed consent (e.g. has intellectual disability)
2. The participant is a paediatric patient (aged below 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Epilepsy Monitoring Unit in Beaumont Hospital who have a history of tonic-clonic seizures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Epilepsy Inventory (QOLIE-31) | Prior to admission